CLINICAL TRIAL: NCT05221437
Title: Personalised Risk Assessment in Febrile Illness to Optimise Real-life Management Across the European Union (PERFORM)
Brief Title: Management and Outcome of Fever in Children in Europe
Acronym: MOFICHE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: REC ref: 16/LO/1684-S
Record Dates: First submitted 2022-01-18; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Antibiotic Prescription

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: antibiotic prescription

SUMMARY:
This is an observational study assessing the management and outcome of children presenting to Emergency Departments (ED) with fever across Europe.

DETAILED DESCRIPTION:
This is an observational study assessing the management and outcome of children presenting to Emergency Departments (ED) with fever across Europe. This study will use large departmental datasets to collect information on at least 50,000 febrile episodes . This study will use large-scale, pseudo-anonymized departmental data, and will not involve consented patient recruitment; nor will it use patient samples. Data included in MOFICHE will be based on that collected as part of routine clinical care. Antibiotic prescription, hospitalisation and number/type of investigations, re-attendance at ED within 5 days of the first hospital presentation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* aged 0- 18 years visiting the emergency care.
* fever measured at ED or history of (measured) fever less than 3 consecutive days prior to presentation at emergency department

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Febrile children aged 0- 18 years visiting the emergency care.
Sampling Method: Non-Probability Sample
Enrollment: 38480 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescription | one year
  number of antibiotic prescriptions
hospitalization | one year
  number of children requiring admission to hospital
Number of investigations | one year
  number of investigations
Number of children re-attending within 5 days of the first hospital presentation. | one year
  Number of re-attendance

IPD SHARING:
Plan to Share IPD: No